CLINICAL TRIAL: NCT02501798
Title: The Effects of Long-acting Methylphenidate on Academic Activity and Related Constructs in Children With ADHD: A Randomised Placebo Controlled Trial
Brief Title: The Effects of Long-acting Methylphenidate on Academic Activity and Related Constructs in Children With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Anne Fleur Kortekaas-Rijlaarsdam, A.F. Kortekaas-Rijlaarsdam, VU University of Amsterdam
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VU-2012-000492-17
Record Dates: First submitted 2014-04-09; First posted 2015-07-17 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Methylphenidate; Academic; Motivation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Methylphenidate (Experimental): Drug: Methylphenidate 7 days dosage as (prior to study) clinically titrated long acting Equasym (brand)
  Interventions: Drug: Methylphenidate
- Drug: Placebo (Active Comparator): Drug: Placebo 7 days Empty green-yellow capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Drug: Methylphenidate
  Other Names: Equasym
  Arms: Drug: Methylphenidate
Drug: Placebo — Drug: Placebo
  Other Names: empty capsule
  Arms: Drug: Placebo

SUMMARY:
This study aims at investigating the direct effects of methylphenidate on school performance of primary school children. Although behavioral effects of this frequently prescribed drug are thoroughly studied (and confirmed), the effects of methylphenidate on school performance are less clear. Recent overviews indicate that effects are mainly quantitative and subject-specific. To gain more insight in this issue, the current double blind placebo controlled crossover study investigates not only the effects of methylphenidate on school performance but also it's effect on related variables such as short term memory, motivation and behavior. 60 children with ADHD are included and tested twice (with medication and with placebo) at their primary school.

DETAILED DESCRIPTION:
Rationale: ADHD (attention deficit hyperactivity disorder) is a common childhood developmental disorder. Besides the behavioural symptoms of ADHD, many children with ADHD experience problems with academic activities. More specifically, these children show problems with math, spelling and reading. The most common treatment for ADHD is medical treatment with methylphenidate (MPH). This treatment is effective in the reduction of ADHD symptoms. However, it is unclear whether treatment with MPH can also improve academic activity. If MPH improves academic activity, it is of great interest to understand which variables influence or mediate this effect. The results from this study can give more insight in the working mechanisms and effectiveness of MPH in reducing the academic problems commonly observed in children with ADHD.

Objectives: The main objective of this study is to assess the impact of MPH on academic activity and to estimate the role of three putative mediators in this relation.

Study design and population: This study is a randomised, double-blind, placebo-controlled cross-over design with a patient group and a control group. Main study parameters/endpoints: The main study parameters are changes in academic activity (ability, effort and engagement). In addition, changes in putative mediators are assessed.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis (DSM-IV)
* primary school education
* sufficient knowledge of Dutch language

Exclusion Criteria:

* neurological or psychiatric disorder other than ODD, CD, learning disorder, dyslexia, anxiety disorder

Healthy volunteers are accepted for the control group

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mathematical performance | 3.5 years
  A standardized task for mathematics is used. Productivity (% completed) and accuracy (%correct) will be calculated for analysis.
Reading performance | 3.5 years
  A standardized task for technical reading ability is used. Productivity (% completed) and accuracy (%correct) will be calculated for analysis.
Spelling performance | 3.5 years
  A standardized task for spelling is used. Productivity (% completed) and accuracy (%correct) will be calculated for analysis.

SECONDARY OUTCOMES:
Cognitive performance | 3.5 years
  Cognitive performance will be measured with standardized tasks for interference control, verbal and spatial working memory. Using principal component analysis a combined (composite) score for cognitive performance will be calculated based on correlations between the measures.
Academic motivation | 3.5 years
  Academic motivation will be measured with a questionnaire measuring intrinsic motivation for schoolwork. In addition, an academic competence questionnaire will be completed by children, parents and teachers separately. A composite score will be calculated of these measures.
Classroom behavior | 3.5 years
  Classroom behavior will be measured with observation scales (by an independent observer) and behavioral rating scales (completed by teachers). Using principal component analysis, these scales will be combined (composite scores), depending on correlations between the measures.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Oosterlaan, Prof. Dr., Principal Investigator — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands